CLINICAL TRIAL: NCT03181607
Title: The 3rd Affiliated Hospital, Guangzhou Medical University
Brief Title: Efficacy and Adverse Effects of Nucleoside Analogues (TDF/LDT) in Preventing Mother-to-child Transmission of HBV
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Xingfei Pan (Other)
Responsible Party: Sponsor-Investigator, Xingfei Pan, Vice Director of Infectious diseases, The Third Affiliated Hospital of Guangzhou Medical University
Organization: The Third Affiliated Hospital of Guangzhou Medical University (Other)
Other Study IDs: [2017] No.157
Record Dates: First submitted 2017-06-02; First posted 2017-06-09 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Chronic Hepatitis b; Women
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mother-to-Child-Transmission (MTCT) of HBV is the most important route in high endemic countries. Although active-passive immune prophylaxis is generally administrated to infants delivered by HBsAg positive women, there are a lot of people infected with HBV in China. High HBV DNA load (>10^5IU/ml) is the vital cause of MTCT. So some researchers used TDF （tenofovir） or LDT（telbivudine） to treat patients with high HBV DNA load during middle, late pregnancy, in order to decrease MTCT. As a result, some data about it were gradually reported in late years. Recently, American Association for the Study of Liver Diseases, European Association for the Study of Liver Diseases and China guidelines for CHB (chronic hepatitis B) suggest that pregnant women with high HBV DNA load be treated with TDF or LDT at 24-28 weeks of gestation to lower MTCT of HBV.

Although TDF or LDT is classified as pregnancy B drugs by FDA, and many studies report that MTCT rate of HBV decreases after women with high HBV DNA load are administrated with TDF or LDT at 24-28 weeks of gestation, a few birth defects are reported. Furthermore, the long-effect of TDF or LDT on infants remains unclear thoroughly.

Some CHB women had severe liver dysfunction before pregnancy or during pregnancy, and routine liver protection therapy could not effect. Some of them could develop into liver failure, fibrosis, cirrhosis, and even died. Moreover, severe liver dysfunction often leads to adverse effects to pregnant women and fetuses, such as pregnancy failure, lower weight, premature birth, etc. As a result, these women have to accept TDF or LDT before pregnancy, or during early pregnancy. So the long-effect of TDF or LDT on infants needs thoroughly investigating.

Taken together, the investigators will enroll women with chronic HBV infection and evaluate their state of illness. Then the investigators treat participants with TDF or LDT or routine liver protection therapy, and follow up the participants for a long period. The investigators' objectives are as follows:

A, To clarify efficacy and adverse effects of TDF/LDT in preventing MTCT between immune-tolerant and immune-active CHB patients.

B, To clarify efficacy and adverse effects of TDF/LDT in preventing MTCT during different trimesters of pregnancy.

C, To compare MTCT rate between patients received TDF/LDT therapy and patients without TDF/LDT therapy.

D, To compare MTCT rate and adverse effects between LDT and TDF.

ELIGIBILITY:
Inclusion Criteria:

* Age of 20-40 years.
* The history of HBV infection ≥6 months.
* Positive for HBsAg.
* For immune-tolerant patients, HBV DNA load of ≥ 10^6IU/ml at 24-28 weeks of gestation.
* For patients already administrated with nucleoside analogues (NA) treatment, the therapy could be not discontinued and TDF or LDT should be used to treat these patients.
* For patients never administrated with NA treatment, ALT ≥2 times of the upper limit of normal (ULN), HBV DNA load of ≥ 10^4IU/ml (positive for HBeAg) or HBV DNA load of ≥ 10^3IU/ml (negative for HBeAg), traditional protecting liver and reducing enzyme treatment was failed.
* The good compliance of patients.

Exclusion Criteria:

* Patients with antibodies against HIV, HCV, HDV, or other forms of chronic liver disease.
* Evidence of hepatocellular carcinoma, decompensated liver disease, auto-immune hepatitis, or significant renal, cardiovascular, respiratory or neurological comorbidity.
* Concurrent treatment with nephrotoxic drugs, glucocorticoids, cytotoxic drugs, nonsteroidal anti-inflammatory drugs, or immune modulators.
* Ultra-sonographic evidence of fetal deformity, abnormal fetal development or placental abnormality.
* Clinical signs of threatened miscarriage.
* History of complication of pregnancy.
* Presence of chronic HBV infection in the biologic father.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Child-bearing age women with chronic HBV infection, who already become pregnant or plan to become pregnant recently,and visit in our hospital, are enrolled.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-05-26 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of hepatitis B infections in the infants at 1 year of age | Between 7-12 months after birth
  Testing for HBsAg in the infants between 7 and 12 months of age

SECONDARY OUTCOMES:
The proportion of birth defects in the infants at 1 month age | From birth to 1 month age
  Measuring the number of infants with congenital abnormality
Growth parameters of the infants | From birth to 5 years age
  The infants'physical development status (head circumference, weight, and height) is measured and analyzed, respectively. Denver Developmental Screening Test is also analyzed.
HBV DNA quantification of mothers | From time of the inclusion to 5 years.
  HBV DNA quantification is detected at 24-28 weeks of gestation, at birth, every 6 month after postpartum.
ALT levels of mothers | From time of the inclusion to 5 years.
  ALT levels are measured every month during pregnancy and the first 3 months postpartum, and every 6 month from the fourth month of postpartum.
HBeAg conversion rate of mothers | From time of the inclusion to 5 years.
  HBeAg quantification is measured every 6 month.

CONTACTS AND LOCATIONS:
Overall Officials: Xingfei Pan, Dr., Study Director — The 3rd Affiliated Hospital, Guangzhou Medical University
Locations (1):
- The 3rd Affiliated Hospital, Guangzhou Medical University, Guanzhou, Guangdong, China